CLINICAL TRIAL: NCT06066697
Title: SOVA Ambassadors Community Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As a result of insufficient remaining funds and the expiration of the project timeline
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ana Radovic, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY23020021; R21MD016143 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Adolescent; Adolescent Medicine; Mental Health Services; eHealth; Online Systems; Primary Healthcare; Social Media; Social Support
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician conducting analyses will be blinded to randomized arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOVA Peer Ambassador Program (Experimental): Participants will be given login information for a website sova.pitt.edu. They will be given weekly emails notifications about new posts. The participant will be onboarded as a blogging peer ambassador. The participant will be expected to contribute content to the website at least once a month by
  1. writing a blog article
  2. sending information (de-identified photo or video or music) to post
     • If they choose this option they will be encouraged to submit their own photo, video, or music to the website or they will be encouraged to write a response to a photo, video, or music piece.
  3. being interviewed by the RA and then the RA "ghostwriting" an article about the interview which they pre-approve prior to it being posted.
  Interventions: Behavioral: SOVA Ambassador
- attention control: brief psychoeducational independent assignments (Active Comparator): Participants will be sent a REDCap form where they will receive a link to a SOVA article to read and a question for them to answer about what they read that will be accessible only to the study team. They will be asked to do this a couple times a month and will be reminded about their participation.
  Interventions: Behavioral: Self-Reflection

INTERVENTIONS:
Behavioral: SOVA Ambassador — The SOVA Ambassador intervention includes:
  adolescents will have access to the website specifically for adolescents: sova.pitt.edu These anonymous websites aim to: (1) challenge negative health beliefs and increase depression/anxiety knowledge through daily blog posts enhanced with peer commentary; (2) promote social support through online peer interactions; and (3) encourage parent-adolescent mental health communication through same day blog posts with questions for discussion.
  Participants that receive this intervention will contribute monthly articles and regular comments.
  Arms: SOVA Peer Ambassador Program
Behavioral: Self-Reflection — Participant will be given an article from the sova.pitt.edu website and a prompt to write about privately.
  Arms: attention control: brief psychoeducational independent assignments

SUMMARY:
The purpose of this study is to examine participant adherence to intervention feasibility and acceptability of intervention, attention control, and implementation strategy.

DETAILED DESCRIPTION:
A 1:1 pilot randomized controlled trial of the SOVA Peer Ambassador Program compared to attention control: brief psychoeducational independent assignments (i.e. reading SOVA articles and responding to open-ended questions without content creation and without peer interaction) (N=40) and evaluate feasibility of implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 to 21

Can read and understand English

Has completed 6th grade

Scores at least 5 or greater on the PHQ-8 (depression) and/or 5 or greater on GAD-7 (anxiety) consistent with at least mild symptoms

Exclusion Criteria:

* no access to internet

Has an intellectual or physical ability which prohibits reading text on the internet (can participate if able to use with assistance, e.g. can use text to speech)

No active email account (can participate if plans to create one)

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Radovic, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Trial outcome data can be accessed by contacting the study principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- SOVA Peer Ambassador Program: Participants will be given login information for a website sova.pitt.edu. They will be given weekly emails notifications about new posts. The participant will be onboarded as a blogging peer ambassador. The participant will be expected to contribute content to the website at least once a month by
  1. writing a blog article
  2. sending information (de-identified photo or video or music) to post
     • If they choose this option they will be encouraged to submit their own photo, video, or music to the website or they will be encouraged to write a response to a photo, video, or music piece.
  3. being interviewed by the RA and then the RA "ghostwriting" an article about the interview which they pre-approve prior to it being posted.
  SOVA Ambassador: The SOVA Ambassador intervention includes:
  adolescents will have access to the website specifically for adolescents: sova.pitt.edu These anonymous websites aim to: (1) challenge negative health beliefs and increase depression/anxiety knowledge through daily blog posts enhanced with peer commentary; (2) promote social support through online peer interactions; and (3) encourage parent-adolescent mental health communication through same day blog posts with questions for discussion.
  Participants that receive this intervention will contribute monthly articles and regular comments.
Period: Overall Study
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Started | 6 | 6
6 Week Completion | 4 | 6
Completed | 1 | 6
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.4) | 15.9 (1.7) | 15.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
MacArthur Scale of Subjective Social Status (National) [Mean (Standard Deviation); unit: units on a scale] — Asked to use a 1 to 10 ladder to rank one's social status as compared to everyone else in the United States; a higher rank indicates a higher social status; the range is 1-10
  units on a scale | 6.1 (2.2) | 5.9 (1.8) | 6.0 (2.0)
Depression Severity [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 measures depression severity a higher score indicating greater severity.
  The PHQ-8 version was used with the 9th item omitted, score range is 0 to 24
  units on a scale | 6.83 (1.60) | 8.83 (2.99) | 7.83 (2.29)
Anxiety Severity [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorders 7-item Questionnaire measures extent of anxiety symptoms. The total score ranges from 0 to 21 with a higher score indicating greater severity.
  units on a scale | 5.67 (2.5) | 7.5 (2.81) | 6.59 (2.65)
Self-Esteem [Mean (Standard Deviation); unit: units on a scale] — The 10-item Rosenberg Self-Esteem Scale (RSES) (α = 0.93) will be administered to assess participants' self-esteem. Scores range from 10-40 with a higher score equating to higher self esteem.
  units on a scale | 28.3 (3.8) | 28.2 (4.4) | 28.3 (3.9)
Emotional Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Emotional self-efficacy will be assessed using The Mental Health Self-Efficacy Scale (MHSES) (α = 0.82). MHSES was developed according to guidelines by Bandura as to how to create self-efficacy questionnaires. The questionnaire contains six items asking about the participant's confidence level in performing mental health self-care behaviors. Scoring of the MHSES is based on a 10-point Likert scale ranging from 1 ("Not at all confident") to 10 ("Totally confident"). Scores are a mean score ranging 1-10 with higher scores meaning higher mental health self-efficacy.
  units on a scale | 6.4 (1.9) | 6.2 (1.4) | 6.3 (1.6)
Social Support [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcome Study Social Support Scale measures types of social support. Higher levels associated with greater support. We will use the emotional/informational subscale from this report and calculate the mean per item score on a range of 1 to 5.
  units on a scale | 3.2 (0.8) | 3.4 (1.0) | 3.3 (0.9)
Social Isolation [Mean (Standard Deviation); unit: units on a scale] — The revised UCLA Loneliness Scale will be administered to all participants to measure social isolation (α = 0.93). This 20-item scale measures one's feelings of social isolation and is scored using a four-point scale (1 = never; 2 = rarely; 3 = sometimes; 4 = often). Score range 20-80, higher score is higher isolation.
  units on a scale | 50.2 (5.6) | 44 (6.6) | 47.1 (6.7)
Stigma [Mean (Standard Deviation); unit: units on a scale] — The Depression Stigma Scale measures stigmatizing attitudes toward depression treatment. It is a continuous measure and the total score ranges from 0-36. There are two subscales: the personal stigma subscale which totals 0-18 and the perceived stigma subscale which totals 0-18. These two are summed for the total stigma score. A higher score indicates a worse outcome.
  units on a scale | 18.8 (6.9) | 19.7 (9.9) | 19.2 (8.1)
Resilience/Positive Youth Development [Mean (Standard Deviation); unit: units on a scale] — Positive Youth Development will be assessed using The Positive Youth Development Very Short Form (PYD-VSF). The confidence subscale is reported which has 3 items with a total score ranging from 3 to 13 (α = 0.78), a higher score associated with a greater level of confidence.
  units on a scale | 8.5 (3.1) | 8.5 (3.0) | 8.5 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: Average number of articles written per participant; Research team extract data from websites and observation notes
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: content pieces
Arm/Group | SOVA Peer Ambassador Program
Number analyzed (Participants) | 6
content pieces | 1.67 (1.75)

2. Secondary Outcome: Feasibility of Control Arm
Description: Average number of submissions to questions on the REDCap form per participant in the Attention control arm Research team extract data from REDCap
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: entries
Arm/Group | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 6
entries | 5.5 (1.2)

3. Secondary Outcome: Acceptability of Intervention
Description: Acceptability of Intervention Measure; Open-ended question (asked the SOVA Website meets my approval)
Time Frame: 12 weeks
Population: 5 individuals in SOVA Ambassador arm did not complete 12 week measure, lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
Participants
  The SOVA website meets my approval.: Completely Agree | 0 | 3
  The SOVA website meets my approval.: Agree | 1 | 3
  The SOVA website meets my approval.: Neither Agree nor Disagree | 0 | 0
  The SOVA website meets my approval.: Disagree | 0 | 0
  The SOVA website meets my approval.: Completely Disagree | 0 | 0
  The SOVA website is appealing to me.: Completely Agree | 0 | 2
  The SOVA website is appealing to me.: Agree | 1 | 4
  The SOVA website is appealing to me.: Neither Agree nor Disagree | 0 | 0
  The SOVA website is appealing to me.: Disagree | 0 | 0
  The SOVA website is appealing to me.: Completely Disagree | 0 | 0
  I like the SOVA website.: Completely Agree | 0 | 2
  I like the SOVA website.: Agree | 1 | 3
  I like the SOVA website.: Neither Agree nor Disagree | 0 | 1
  I like the SOVA website.: Disagree | 0 | 0
  I like the SOVA website.: Completely Disagree | 0 | 0
  I welcome the SOVA website.: Completely Agree | 0 | 2
  I welcome the SOVA website.: Agree | 1 | 4
  I welcome the SOVA website.: Neither Agree nor Disagree | 0 | 0
  I welcome the SOVA website.: Disagree | 0 | 0
  I welcome the SOVA website.: Completely Disagree | 0 | 0

4. Secondary Outcome: Acceptability of Implementation Strategy
Description: Open-ended question: How acceptable to you was it to participate in this program? (referring to mental health program used as an implementation strategy) asked at baseline
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 6 | 6
Participants
  Very acceptable | 3 | 3
  Somewhat acceptable | 0 | 0
  Neither | 1 | 0
  Somewhat unacceptable | 0 | 0
  Very unacceptable | 0 | 0
  Did not attend program | 2 | 3

5. Secondary Outcome: Acceptability of Randomization
Description: Single item open-ended question inquiring how acceptable it was to being randomly chosen to participate in the SOVA Ambassador arm versus the control arm
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
Participants
  Very Acceptable | 0 | 3
  Somewhat Acceptable | 1 | 3
  Neither | 0 | 0
  Somewhat Unacceptable | 0 | 0
  Very Unacceptable | 0 | 0

6. Secondary Outcome: Depression Severity
Description: Patient Health Questionnaire-9 measures depression severity a higher score indicating greater severity.
  The PHQ-8 version was used with the 9th item omitted, score range is 0 to 24
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 9.00 (6.68) | 9.50 (3.02)

7. Secondary Outcome: Depression Severity
Description: as for outcome 6
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 9 (NA) — Standard Deviation not calculable for one participant | 8 (5.4)

8. Secondary Outcome: Anxiety Severity
Description: Generalized Anxiety Disorders 7-item Questionnaire measures extent of anxiety symptoms. The total score ranges from 0 to 21 with a higher score indicating greater severity.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 7.5 (6.24) | 7.5 (3.08)

9. Secondary Outcome: Anxiety Severity
Description: as for outcome 8
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 7 (NA) — Standard Deviation not calculable for one participant | 5.5 (2.88)

10. Secondary Outcome: Resilience/Positive Youth Development
Description: Positive Youth Development will be assessed using The Positive Youth Development Very Short Form (PYD-VSF). The confidence subscale is reported which has 3 items with a total score ranging from 3 to 13 (α = 0.78), a higher score associated with a greater level of confidence.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 7 (2.3) | 8.7 (2.3)

11. Secondary Outcome: Resilience/Positive Youth Development
Description: as for outcome 10
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 4 (NA) — Standard Deviation not calculable for one participant | 7.8 (1.9)

12. Secondary Outcome: Self-Esteem
Description: The 10-item Rosenberg Self-Esteem Scale (RSES) (α = 0.93) will be administered to assess participants' self-esteem. Items on the Rosenberg Self-Esteem Scale ask about self-worth and self-acceptance and are scored using a four-point scale from 1 = strongly disagree, to 4 = strongly agree. The scores on each question are summed together, with higher scores indicating greater self-esteem. Scores range from 10-40 with a higher score equating to higher self esteem.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 26.0 (3.7) | 26.3 (2.2)

13. Secondary Outcome: Self-Esteem
Description: The 10-item Rosenberg Self-Esteem Scale (RSES) (α = 0.93) will be administered to assess participants' self-esteem. Items on the Rosenberg Self-Esteem Scale ask about self-worth and self-acceptance and are scored using a four-point scale from 1 = strongly disagree, to 4 = strongly agree. The scores on each question are summed together, with higher scores indicating greater self-esteem. Scores range from 10-40
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
score on a scale | 25 (NA) — Standard Deviation not calculable for one participant | 28.8 (5.7)

14. Secondary Outcome: Emotional Self-Efficacy
Description: Emotional self-efficacy will be assessed using The Mental Health Self-Efficacy Scale (MHSES) (α = 0.82) Clarke 2014. MHSES was developed according to guidelines by Bandura as to how to create self-efficacy questionnaires (Bandura, 2006) . The questionnaire contains six items asking about the participant's confidence level in performing mental health self-care behaviors. Scoring of the MHSES is based on a 10-point Likert scale ranging from 1 ("Not at all confident") to 10 ("Totally confident"). Scores are a mean score ranging 1-10 with higher scores meaning higher mental health self-efficacy.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 6.7 (0.9) | 6.3 (1.0)

15. Secondary Outcome: Emotional Self-Efficacy
Description: as for outcome 14
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 6 (NA) — Standard Deviation not calculable for one participant | 7.3 (1.5)

16. Secondary Outcome: Social Support
Description: The Medical Outcome Study Social Support Scale measures types of social support. Higher levels associated with greater support. We will use the emotional/informational subscale from this report and calculate the mean per item score on a range of 1 to 5.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 3.3 (0.7) | 3.1 (0.3)

17. Secondary Outcome: Social Support
Description: as for outcome 16
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 3.6 (NA) — Standard Deviation not calculable for one participant | 3.2 (0.8)

18. Secondary Outcome: Social Isolation
Description: The revised UCLA Loneliness Scale will be administered to all participants to measure social isolation (α = 0.93). This 20-item scale measures one's feelings of social isolation and is scored using a four-point scale (1 = never; 2 = rarely; 3 = sometimes; 4 = often) . Score range 20-80, higher score is higher isolation.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 52 (8.6) | 42.2 (4.8)

19. Secondary Outcome: Social Isolation
Description: as for outcome 18
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 50 (NA) — Standard Deviation not calculable for one participant | 40.7 (8.4)

20. Secondary Outcome: Stigma
Description: The Depression Stigma Scale measures stigmatizing attitudes toward depression treatment. It is a continuous measure and the total score ranges from 0-36. There are two subscales: the personal stigma subscale which totals 0-18 and the perceived stigma subscale which totals 0-18. These two are summed for the total stigma score. A higher score indicates a worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 4 | 6
units on a scale | 19.8 (3.9) | 18.5 (2.3)

21. Secondary Outcome: Stigma
Description: as for outcome 20
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
Number analyzed (Participants) | 1 | 6
units on a scale | 12 (NA) — Standard Deviation not calculable for one participant | 17.0 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the time period of the study participant enrollment (12 weeks)
Arm/Group | SOVA Peer Ambassador Program | Attention Control: Brief Psychoeducational Independent Assignments
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
All collected data for pre-specified primary and secondary outcome measures were summarized and reported in the outcome measure data tables. The planned statistical analyses were not performed due to insufficient enrollment and additional pre-planned analyses being statistically inappropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT06066697/Prot_SAP_002.pdf
  • Informed Consent Form (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT06066697/ICF_003.pdf